CLINICAL TRIAL: NCT03774030
Title: Evaluation and Optimization of Hearing Devices in 3-D Complex Audio Environments Study 2
Acronym: HEAR3D_CE2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sonova AG (Industry)
Collaborators: Swiss Commission for Technology and Innovation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2017-02051-2
Record Dates: First submitted 2018-12-11; First posted 2018-12-12 (Actual); Last update posted 2019-05-09 (Actual); Status verified 2019-05

CONDITIONS: Ability, Spatial
MeSH Terms: conditions — Spatial Navigation

STUDY DESIGN:
Intervention Model Description: a group of hearing-impaired particpants with mild or severe hearing loss
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- hearing impaired participants (Experimental): Hearing impaired participants with mild or severe hearing loss
  Interventions: Procedure: several virtual 3-D complex audio environments

INTERVENTIONS:
Procedure: several virtual 3-D complex audio environments — The focus is a comparison of 3 hearing aid algorithms in a virtual 3-D complex audio Environment.

SUMMARY:
A methodical evaluation of novel sound changing principles in CE-labelled Sonova brand hearing instruments (e.g. Phonak hearing instruments) is intended to be conducted on hearing impaired participants. These sound changing principles are enabled by respective hearing instrument technologies and hearing instrument algorithms. The aim of the study is to investigate and assess strengths and weaknesses of these novel sound changing principles in terms of hearing performance to determine their application in hearing instruments (Phase of development). Both, objective laboratory measurements as well as subjective evaluations in real life environment will be carried out. This will be a controlled, single blinded and randomised active comparator clinical evaluation which will be conducted mono centric at the University Hospital of Zürich.

ELIGIBILITY:
Inclusion Criteria:

* Adult persons (minimum age: 18 years) with Hearing loss
* Healthy outer ear (without previous surgical procedures)
* Ability to fill in a questionnaire conscientiously
* Informed Consent as documented by signature

Exclusion Criteria:

* Contraindications to the MD in this study, e.g. known hypersensitivity or allergy to the investigational product
* Limited mobility and not in the position to attend weekly appointments
* Limited ability to describe listening impressions/experiences and the use of the hearing aid
* Inability to produce a reliable hearing test result
* Massively limited dexterity
* Known psychological problems
* Known central hearing disorders

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-10-09 (Actual); Primary Completion 2019-01-21 (Actual); Study Completion 2019-01-21 (Actual)

PRIMARY OUTCOMES:
Head movements measured with head tracker | 6 weeks
  The participant starts the acoustic stimulus, tries to identify the direction of the stimulus as precise as possible and validates the final position. This is interpreted as reaction time with regard to spatial quality in seconds [s].

CONTACTS AND LOCATIONS:
Overall Officials: Norbert Dillier, Professor, Principal Investigator — University Hospital
Locations (1):
- University Hospital Zurich, Zurich, Switzerland

REFERENCES:
- [Result] Gatehouse S, Noble W. The Speech, Spatial and Qualities of Hearing Scale (SSQ). Int J Audiol. 2004 Feb;43(2):85-99. doi: 10.1080/14992020400050014. PMID 15035561
- [Result] Choisel S, Wickelmaier F. Evaluation of multichannel reproduced sound: scaling auditory attributes underlying listener preference. J Acoust Soc Am. 2007 Jan;121(1):388-400. doi: 10.1121/1.2385043. PMID 17297794
- [Result] Mueller MF, Meisenbacher K, Lai WK, Dillier N. Sound localization with bilateral cochlear implants in noise: how much do head movements contribute to localization? Cochlear Implants Int. 2014 Jan;15(1):36-42. doi: 10.1179/1754762813Y.0000000040. Epub 2013 Nov 25. PMID 23684420
- [Result] Catic J, Santurette S, Dau T. The role of reverberation-related binaural cues in the externalization of speech. J Acoust Soc Am. 2015 Aug;138(2):1154-67. doi: 10.1121/1.4928132. PMID 26328729
- [Result] Simon LS, Zacharov N, Katz BF. Perceptual attributes for the comparison of head-related transfer functions. J Acoust Soc Am. 2016 Nov;140(5):3623. doi: 10.1121/1.4966115. PMID 27908072
- See also: link to first part of study — https://clinicaltrials.gov/ct2/show/NCT03514758?term=sonova&draw=3&rank=21